CLINICAL TRIAL: NCT07157163
Title: Effectiveness of Nudge and Motivational Interviewing Interventions to Improve Influenza Vaccination Uptake Among Healthcare Workers in China: a Two-phase Randomized Controlled Trial
Brief Title: Nudge and Motivational Interviewing Interventions to Improve Influenza Vaccine Uptake Among Healthcare Workers in China
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centers for Disease Control and Prevention, China (Other Government)
Responsible Party: Principal Investigator, Lixin Hao, Chief Physician of National Immunization Program, Centers for Disease Control and Prevention, China
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 202529
Record Dates: First submitted 2025-08-19; First posted 2025-09-05 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Influenza Vaccine; Healthcare Workers
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Data analysts
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Phase 1: standardized nudge group (Experimental): Participants receive uniform nudge messages.
  Interventions: Behavioral: Phase 1: standardized nudge messages
- Phase 1: personalized nudge group (Experimental): Participants receive tailored nudge messages with access to a chatbot.
  Interventions: Behavioral: Phase 1: personalized nudge messages + chatbot
- Phase 1: control group (No Intervention): Participants receive no study-related interventions.
- Phase 2: motivational interviewing group (Experimental): Participants receive motivational interviewing.
  Interventions: Behavioral: Phase 2: motivational Interviewing
- Phase 2: control group (No Intervention): Participants receive no study-related interventions.

INTERVENTIONS:
Behavioral: Phase 1: standardized nudge messages — Participants receive uniform messages designed to encourage influenza vaccination. These messages, grounded in nudge theory, are delivered through a Chinese online platform to promote vaccination uptake.
  Arms: Phase 1: standardized nudge group
Behavioral: Phase 1: personalized nudge messages + chatbot — Participants receive tailored messages designed to encourage influenza vaccination. These messages, grounded in nudge theory, are delivered through a Chinese online platform to promote vaccination uptake. Additionally, they have access to an interactive chatbot to address questions and provide decision-making support for influenza vaccination.
  Arms: Phase 1: personalized nudge group
Behavioral: Phase 2: motivational Interviewing — Unvaccinated participants engage in one-on-one motivational interviewing sessions with a trained interviewer.
  Arms: Phase 2: motivational interviewing group

SUMMARY:
The goal of this clinical trial is to learn if nudge-based interventions and motivational interviewing work to improve influenza vaccination uptake among healthcare workers in China. A two-phase randomized controlled trial will be conducted in community hospitals across China, targeting healthcare workers as participants.

The main questions are:

Do nudge-based interventions increase vaccination rates among healthcare workers?

Does motivational interviewing increase vaccination compliance among those who remain unvaccinated after the phase 1?

In phase 1, community hospitals will be randomized as units into three arms: standard nudge group, personalized nudge group, and a control group. In phase 2, healthcare workers who remain unvaccinated after phase 1 will be individually randomized to either a motivational interviewing group or a control group.

Participants will:

Be recruited from community hospitals to participate in the study. In phase 1 (at the early stage of the flu season), community hospitals will be randomly assigned to one of three groups: standardized nudge messages, personalized nudge messages with a chatbot, or no reminders.

If still unvaccinated in phase 2 (during peak flu season), healthcare workers will be individually assigned to either motivational interviewing group or receive no extra contact.

Have their vaccination status checked at the end of each phase.

DETAILED DESCRIPTION:
A two-phase randomized controlled trial will be conducted to evaluate the effectiveness of multi-component interventions to improve vaccination uptake, targeting healthcare workers in China.

Sample size Phase 1: Cluster-Randomized Controlled Trial The sample size is determined to identify a significant difference in the primary outcome, defined as the influenza vaccination uptake among healthcare workers in community hospital, comparing the intervention and control groups. Historical surveillance data from the three participating cities indicate a baseline vaccination rate of approximately 4% without targeted interventions. The proposed intervention is expected to increase this rate to 10%. A two-sided significance level of α = 0.05 is set, adjusted to α = 0.0167 via Bonferroni correction to account for three planned pairwise comparisons. Statistical power is set at 0.80, with an assumed intraclass correlation coefficient (ICC) of 0.05 and an average cluster size of 50 participants per cluster. Based on these parameters, 23 clusters per study arm are required, resulting in a total of 69 clusters across the three arms. To account for potential attrition, the sample size will be increased to 27 clusters per arm, yielding a total of 81 clusters and an estimated 4,050 participants. All eligible healthcare workers in the participating community hospitals will be included in the study.

Phase 2: Individual Randomized Controlled Trial In phase 2, the target population comprises healthcare workers who remain unvaccinated after Phase 1, from the 54 community hospitals assigned to the intervention arms. Without further intervention, the vaccination uptake rate in this group is estimated to be approximately 3%. The motivational interviewing intervention is expected to increase this rate to 13%. Assuming a two-sided significance level of α = 0.05 and statistical power of 0.80, sample size estimation indicates a minimum of 112 participants per group is required. To ensure feasibility and maintain study power, the motivational interviewing group will aim to enroll 150 participants. Fifteen community hospitals will be randomly selected from the two intervention arms of Phase 1. Control groups are established: 1) healthcare workers from 15 community hospitals selected for the motivational interviewing intervention, excluding approximately 10 individuals per community hospital who receive the intervention, resulting in a control group of approximately 525 healthcare workers; and 2) healthcare workers from the remaining 39 community hospitals not participating in the motivational interviewing intervention, comprising approximately 1,755 individuals. Therefore, the control group in phase 2 comprises approximately 2,280 participants.

In phase 1, a stratified block randomization method will be employed to ensure balanced allocation across study groups. Stratification factors include historical influenza vaccination rates among healthcare workers and the size of the healthcare staff at each community hospital. Community hospitals with comparable levels of these factors are grouped into blocks within each city and then randomly assigned within each block to one of three groups: the standardized nudge group, personalized nudge group, or a control group.

In phase 2, a two-stage random sampling procedure will be used. Specifically, 15 community hospitals will be randomly selected from the 54 hospitals assigned to the intervention groups in the phase 1 (five hospitals per province). Within each selected hospital, 10 healthcare workers who remained unvaccinated after the first-phase intervention will be randomly sampled and enrolled in the individual-level intervention study.

Qualitative interviews and a baseline survey will be conducted before the interventions. Follow-up questionnaires will be completed two weeks after the end of each intervention phase. The primary outcome is the receipt of influenza vaccination by healthcare workers, which will be assessed two months after each intervention phase using official vaccination records.

The intention-to-treat (ITT) analysis will be used to evaluate the effectiveness of the interventions. The primary outcome is influenza vaccine uptake among healthcare workers post-intervention. Vaccine uptake will be compared between intervention and control groups, and across intervention arms, using chi-square tests. To account for clustering and adjust for potential confounders, generalized estimating equation (GEE) models will be employed to provide robust effect estimates. Timing of vaccination will be evaluated using Kaplan-Meier survival curves and log-rank tests, with Cox proportional hazards models to estimate intervention effects on time-to-vaccination. Subgroup analyses will assess heterogeneity of intervention effects across populations stratified by baseline characteristics.

Secondary outcomes will be evaluated at baseline and post-intervention. Between-group comparisons, including intervention versus control and across intervention arms, will use t-tests for continuous variables and chi-square tests for categorical variables. GEE models with repeated measures will assess intervention effects on secondary outcomes, adjusting for relevant covariates. Subgroup analyses will examine differential effects across subpopulations defined by baseline factors.

ELIGIBILITY:
Phase 1: Cluster-Randomized Controlled Trial

Inclusion Criteria:

* Full-time employees of community hospitals who remain employed throughout the study period.
* Have not scheduled or received an influenza vaccine between August 2024 and the time of formal enrollment.
* Agree to participate and provide informed consent.

Exclusion Criteria:

* Participants with medical conditions that contraindicate influenza vaccination.
* Participants who refuse to participate or do not provide informed consent .

Phase 2: Individual Randomized Controlled Trial

Inclusion Criteria:

* Healthcare workers from community hospitals who remain unvaccinated after Phase 1, as verified by official records, will be screened.
* A selected subset of these individuals will be invited to participate in Phase 2.

Exclusion Criteria:

- Participants who refuse to participate or do not provide informed consent .

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4050 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Influenza vaccination uptake | 2 months post-intervention for each study phase.
  whether participants get vaccinated against influenza, measured by official vaccination system

SECONDARY OUTCOMES:
Influenza vaccine literacy | Baseline (pre-intervention) and 2 weeks after each intervention phase.
  A series of questions about influenza vaccine knowledge and misinformation. Total literacy score is calculated based on the number of questions answered correctly by the participants.
Influenza vaccine confidence | Baseline (pre-intervention) and 2 weeks after each intervention phase.
  Vaccine confidence index (VCI), including participants' confidence in the importance, effectiveness, and safety of the influenza vaccine, and trust in public health agency. Responses will be measured using a 5-point Likert scale (1 = strongly disagree, 5 = strongly agree).
High perception on influenza risk | Baseline (pre-intervention) and 2 weeks after each intervention phase.
  Proportion of participants who perceived to be susceptible and severe to influenza.
Influenza vaccination intention | Baseline (pre-intervention) and 2 weeks after each intervention phase.
  Participants' intention to receive influenza vaccine. Unit of Measure: Influenza Vaccination Intention 5-point Likert scale score, 1-5 (higher scores indicate stronger intention).
Recommendation of influenza vaccine to the public. | Baseline (pre-intervention) and 2 weeks after each intervention phase.
  Recommendation frequency of influenza vaccine to the public during the health care. Unit of Measure:Recommendation frequency score, 1-5 (higher scores indicate more frequent recommendations).
Access to professional information of influenza vaccine | Baseline (pre-intervention) and 2 weeks after each intervention phase.
  Whether professional information about influenza vaccine is provided in the workplace.

OTHER OUTCOMES:
Intervention usability assessment | 2 weeks after each intervention phase.
  A series of questions assessing usability and feasibility of the interventions.
Cost of interventions | Immediately after the completion of each intervention phase.
  The cost of designing and implementing interventions. Unit of Measure: Chinese Yuan (CNY).

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared due to participant privacy concerns and institutional data protection policies.